CLINICAL TRIAL: NCT01439477
Title: StrongWomen- Healthy Hearts: A Community Based Program for Midlife and Older Women
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Sara C. Folta, Assistant Professor, Tufts University
Other Study IDs: TuftsU-9289
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Overweight and Obesity
Keywords: exercise; healthy eating; heart disease; prevention & control; Middle aged; Women; Health promotion
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity; Motor Activity; Heart Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death for women in the United States. CVD disproportionately affects underserved populations, specifically low-income, minority, and rural women who have higher obesity rates and experience other health disparities. There is a need for replicable, evidence-based programs that target women, particularly midlife and older women who represent an increasing proportion of the U.S. population, to reduce their CVD risk . StrongWomen - Healthy Hearts is a 12-week, community-based program that has demonstrated effectiveness at improving CVD risk factors, including body weight, diet quality, and physical activity in a controlled, randomized trial conducted with midlife and older overweight and obese subjects in Arkansas and Kansas.

The central objective is to rigorously evaluate dissemination of the StrongWomen - Healthy Hearts Program using the RE-AIM framework to achieve maximal public health impact. Expanded dissemination will occur through the Cooperative State Research, Education and Extension Service (CSREES) This partnership will leverage a long and successful collaboration between Tufts University and CSREES that provides strength training programs to older women in 41 states.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 40 years of age
* Female
* BMI greater than 24
* sedentary (not doing any type of exercise more than once per week)

Exclusion Criteria:

* unstable medical condition that would preclude participation in an exercise program
* current participation in another lifestyle modification program
* cognitive impairment
* pregnancy.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women greater than 40 years old who are overweight or obese and sedentary
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Body Weight | 9/2014-7/2015

SECONDARY OUTCOMES:
Waist circumference | 9/2014-7/2015
Percent Body Fat | 9/2014-7/2015
Diet (24-hour recall) | 9/2014-7/2015
Physical Activity (IPAQ) | 9/2014-7/2015
Physical Activity (accelerometer) | 9/2014-7/2015
Cardiorespiratory Fitness (1-Mile Walk Test) | 9/2014-7/2015
Blood Pressure | 9/2014-7/2015
Self-Regulation | 9/2014-7/2015
Collective Efficacy | 9/2014-7/2015
Perceived Stress | 9/2014-7/2015
Self-Efficacy | 9/2014-7/2015
Perceived Social Support | 9/2014-7/2015
Civic Engagement | 9/2014-7/2015

OTHER OUTCOMES:
Adherence | 9/2014-7/2015
Retention | 9/2014-7/2015
Satisfaction with Intervention | 4/2014-7/2015